CLINICAL TRIAL: NCT05409963
Title: Tobacco Impact on Quality of Life, a Cross-sectional Study on Snus-use, Dual Use, Smoke Use and Non-using.
Brief Title: Tobacco Impact on Quality of Life on Snus-use, Dual Use, Smoke Use and Non-using.
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Solbrith Wachsmann, Specialist nurse, phil,mag, Vastra Gotaland Region
Other Study IDs: 65381
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Tobacco Use
Keywords: Cigarette smoking; Health; Population characteristics; Quality of life; Tobacco smokeless.
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study was to compare HRQOL in snus-users and dual users (snus and smoking) with never tobacco users. Secondary aim included comparing HRQOL in smokers with non-smokers.

DETAILED DESCRIPTION:
Tobacco use is a major public health issue. The number of smokers decrease simultaneously as oral moist snuff (called "snus"), is promoted as a healthier alternative in spite its' negative health effects. Studies of health-related quality of life (HRQOL) of those who use snuff are lacking. Recruitment of 674 women and 605 men aged 18 to 65 years through a Swedish population data-base was performed for this cross-sectional study in southwestern Sweden. Subjects completed a questionnaire about tobacco use and the 36-item Short Form Health Survey (SF-36). The non-parametric Mann-Whitney test was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 65 years

Exclusion Criteria:

not understand the Swedish language

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Three thousand women and men were randomly selected by the Swedish population data-base (SPAR) in rural areas of southwest Sweden.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2014-03-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life was measured using SF-36. | The time when the data entry is made, about 8 weeks
  The SF-36 collected data on perceived health status in eight domains: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE) and mental health (MH). The physical component summary (PCS) and mental component summary (MCS). Scores range from 0 to 100 with higher scores representing a higher perceived health
Tobacco habits. | The time when the data entry is made, about 8 weeks
  The term pack-year (numbers of cigarettes / day * number of years / 20) and box-year (numbers of snuff boxes / week * number of years) was used to describe tobacco use. The variables smoking and snuff use were transformed from one pack-year to pack-decades by dividing pack-year by 10. Similarly, box-years were transformed to box-decades and age from years to decades.

CONTACTS AND LOCATIONS:
Overall Officials: Solbrith Wachsmann, DMPhil, Study Director — Region Västra Götaland, Research, Education, Development & Innovation, Primary Care Research, Sweden; Gun Rembeck, PHD, Principal Investigator — Region Västra Götaland, Research, Education, Development & Innovation, Primary Care Research, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wachsmann S, Nordeman L, Billhult A, Rembeck G. Tobacco impact on quality of life, a cross-sectional study of smokers, snuff-users and non-users of tobacco. BMC Public Health. 2023 May 15;23(1):886. doi: 10.1186/s12889-023-15844-z. PMID 37189128